CLINICAL TRIAL: NCT06878820
Title: Nurses in the Lead - Nursing Leadership and Autonomy in Function Focused Care in Hospital: a Prospective Before-after Study
Brief Title: Nurses in the Lead - Nursing Leadership and Autonomy in Function Focused Care in Hospital
Status: Enrolling by invitation | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Collaborators: Erasmus Medical Center (Other); Slingeland Hospital (Other)
Responsible Party: Principal Investigator, jmman, Associate professor, Leiden University Medical Center
Other Study IDs: 134718; 10040022230013 (Other Grant/Funding Number: ZonMw)
Record Dates: First submitted 2024-11-22; First posted 2025-03-17 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Nurse-Patient Relations; Implementation Research; Physical Inactivity; Physical Activities; ADL; Mobility and Independence; Leadership; Interprofessional Team Collaboration; Hospital Care
Keywords: function focused care; implementation; leadership; mobility; ADL; nurses in the lead; nursing care
MeSH Terms: conditions — Sedentary Behavior; Motor Activity | interventions — Hospitals

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Function Focused Care: Nurses provide care according to Function Focused Care in Hospital (FFCiH) principles. After implementation of this intervention, all patients admitted to the selected wards in the hospital receive FFCiH.
  Interventions: Behavioral: Function Focused Care
- Usual Care: Before implementation of Function Focused Care in Hospital, nurses provide care as usual to patients admitted to the selected wards in hospital

INTERVENTIONS:
Behavioral: Function Focused Care — FFCiH is an effective nursing approach and focuses on stimulating nurses to promote patients' self-reliance in daily functioning, encouraging the patients' engagement in daily activities and helping patients to attain and maintain their highest level of function and to increase time spent in physical activity.
  Other Names: FFC; FFCiH; Function Focused Care in Hospital
  Groups: Function Focused Care

SUMMARY:
The goal of this prospective before-after study (observational) is to implement Function Focused Care in Hospital (FFCiH), paying specific attention to the role of nurses and how they can take the leadership and autonomy in the interprofessional collaboration regarding FFCiH. To reach this aim, the researchers defined two sub-objectives:

1. to identify barriers and facilitators (determinants) for nursing autonomy and leadership and application FFCiH in the interprofessional collaboration on a surgical and internal medicine ward to design a tailored implementation strategy for FFCiH. 2. to evaluate the effectiveness of the implementation strategy on nursing leadership and the application of FFCiH.

The investigators developed two work packages related to the two sub-objectives: identifying determinants and strategies for the successful application of FFCiH and nurse leadership, among others, by introducing nurse champions and evaluating their effect on the application of FFCiH. The primary endpoint is the level of application of FFCiH as reflected in adherence to and coverage of FFCiH in daily nursing care.

The secondary endpoints are: 1) for nurses: the nurses' role development with regards to leadership and autonomy in the application of FFCiH by ward nurses and nurse champions, leadership competencies of ward nurses, and autonomy of ward nurses and 2) for patients: physical functioning and independency in mobility and ADL.

Researchers will compare FFCiH with usual care to see if there are differences regarding the outcome measurements.

The study population consists of nurses, physiotherapists, doctors, other member of the interprofessional team, hospitalized patients and their relatives.

Intervention: FFCiH focuses on stimulating nurses to promote patients' self-reliance in daily functioning, encouraging the patients' engagement in daily activities and, helping patients to attain and maintain their highest level of function and increasing time spent in physical activity. FFCiH is a proven effective approach for promoting patients' physical functioning and mobility.

DETAILED DESCRIPTION:
The investigators will conduct a prospective before-after multicenter study, including a process evaluation, with a mixed methods approach in two university medical centers. In the preparation phase before the before-after study the tailored implementation strategy for FFCiH will be developed. Between the before and after phases of the study, the investigators will implement in two or three cyclic processes the FFCiH approach by strengthening nursing leadership and autonomy in the application of FFCiH in the interprofessional collaboration, using the predefined tailored implementation strategy.

ELIGIBILITY:
Nurses and student nurses (vocational nursing educational level (MBO)/ (bachelor nursing educational level (HBO)):

Inclusion Criteria:

- All (student-)nurses working in the participating wards are expected to be involved in application of FFC and role development with regards to leadership and autonomy of nurses and therefore considered to be eligible for participation in the study.

Exclusion Criteria:

- No exclusion criteria were defined for nurses and student nurses.

Physiotherapists, doctors and other member of the interprofessional team;

Inclusion Criteria:

- All professional groups that are part of the interprofessional team of the ward and who work in the participating wards are expected to collaborate with the nursing in their daily care and therefore considered to be eligible for participation in this study.

Exclusion Criteria:

- No exclusion criteria were defined for physiotherapists, doctors and other members of the interprofessional team.

Patients and informal caregivers:

Inclusion Criteria:

- All patients admitted to the participating wards of the 2 hospitals receiving care either before or after the implementation of FFC and the patients informal caregiver as determined by the patient.

Exclusion Criteria:

* A life-threatening situation or in a terminal phase upon admission (only applicable to patients)
* Not mastering the Dutch language;
* Not able to communicate adequately, based on a below threshold score on the MOCA or the FAST (only applicable to patients)
* A second hospitalization on one of the participating wards after being included in the study during the study period;
* An hospitalization < 48 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The domain of this study consists of
  * nurses, physiotherapists, doctors, other member of the interprofessional team (e.g. occupational therapist),
  * patients admitted to a surgical respectively internal medicine ward of a hospital, and their informal caregivers.
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2025-05-05 (Estimated); Study Completion 2025-06-05 (Estimated)

PRIMARY OUTCOMES:
Level of leadership using the Leadership Practices Inventory (LPI) - Nurses | up to four weeks directly before implementation & up to four weeks directly after implementation
  The LPI questionnaire consist of 30 leadership behaviors presented as behavioral statements, that can categorized into 5 subscales, representing five leadership practices: 1) Model the way, 2) Inspire a shared vision, 3) Challenge the process, 4) Enable others to act, and 5) Encourage the heart. Each of these statement can be scored on a 10-point Likert scale, for which a higher score indicate more frequent the respondent engage in the leadership behavior. The internal reliability of the LPI in nurses ranges from 0.66 to 0.96.36 The original questionnaire has been translated into Dutch.
Level of autonomy - Nurses | up to four weeks directly before implementation & up to four weeks directly after implementation
  Using the Maastricht Autonomy Questionnaire (MAQ), which consists of 10 items scored on a five-point Likert scale ranging from very little to very much.The total score ranges from 10 to 50. Higher scores indicate more job autonomy. The questionnaire includes information on job control and freedom in work tasks and methods. It measures the opportunity for staff to determine a variety of task elements, such as the pace of work and the work goals. A sample item is: 'My work offers me the opportunity to interrupt my job whenever I want.' Current study findings confirmed good internal consistency (Cronbach's alpha=0.90).

SECONDARY OUTCOMES:
Adherence (fidelity) | up to four weeks after implementation
  Refers to the extent to which FFCiH has been applied as intended, and will be measured with the key components of FFCiH, such as goal setting with patient, individualized care plan, encouragement of patient's active involvement in ADL and evaluation the level of the patient's ADL-independence and mobility.
  This outcome will be measured with
  1. qualitative focus group interviews with the multidisciplinary team and individual interviews with patients. Topics include the key components of FFCiH.
  2. Screening of electronic patient records. The electronic patient records will be screened on the number of reported short- and long-term goals and the amount of nursing report that contains information about bathing, dressing, mobility or transfers.
Level of mobility - Patients | <72 hours after hospital admission and at discharge (assessed up to 3 days)
  Measured using the AMEXO. this measure is the Amsterdam UMC extension of the John Hopkins Highest Level of Mobility (AMEXO) scale. The instrument consist of twelve categories representing the highest level of mobility. The response categories includes: 1= bed lying; 2= bed turn self/activity; 3= bed sit at edge; 4= chair transfer; 5= stand 1 minute; 6=walk 10+ steps; 7=walk 25+ feet; 8=walk 250+ feet ,9= 225m; 10= 450m; 11= 750m; 12= 1125m.:.'. The higher the total score, the higher the level of independence.
Level of independence in Activities of Daily Livings - patients | <72 hours after hospital admission and at discharge (assessed up to 3 days)
  Measured with the KATZ-ADL. This measurement consists of 6 items: bathing, dressing, toilet visit, movement inside the house, continence, feeding. The items score on a 2 point scale: dependent or independent.
Level of coverage (reach) | up to four weeks after implementation
  Refers to the extent to which patients actually receive FFCiH, and measured by determining the extent to which patients who qualify for FFCiH actually receive it.
  This outcome will be measured with 1) qualitative focus group interviews with the multidisciplinary team and individual interviews with patients. Topics include the key components of FFCiH. 2) Screening of electronic patient records. The electronic patient records will be screened on the number of reported short- and long-term goals and the amount of nursing report that contains information about bathing, dressing, mobility or transfers.
Numbers of days stayed in the hospital - patients | At discharge (assessed up to 14 days)
  Based on the findings in our previous study and known from clinical practice, we know that discharge from hospital highly depends on independence in ADL and/or mobility. As a result, it is expected that a recovery of independence in ADL and mobility primarily does not lead to higher levels of independence in ADL and mobility at discharge, but to a shorter admission with the same level of independence in ADL and mobility. Therefore, we also will collect data from patient files regarding the duration of hospital admission.

OTHER OUTCOMES:
Baseline characteristics nurses | Up to four weeks before implementation
  * age (years)
  * Gender (male, female, other)
  * type of ward of (primarily) employment (surgical, internal medicine, orthopedic surgical, pulmonary, etc.)
  * level of education level (MBO, HBO, Master, PhD)
  * years of experience as health care professional (years)
  * team longevity (years of membership of the team)
Baseline characteristics patients and their informal caregivers | <72 hours after hospital admission
  * Age (years)
  * Gender (male, female, other)
  * educational level (numbers of years of education / last occupation)
  * marital status (single, married/cohabiting, widowed/divorced)
  * living accommodation (independent alone, independent with informal caregiver, independent with others, nursing home)
  * (number of) somatic diagnoses, admission diagnose, (patient)
  * use of walking aid/device (yes/no) (patient)
  * relationship to patient (spouse/partner, child, parent, neighbour, friend) (informal caregiver)

CONTACTS AND LOCATIONS:
Overall Officials: Janneke M de Man - van Ginkel, Principal Investigator — Leiden University Medical Center
Locations (3):
- Netherlands (3):
  - Stichting Slingeland Ziekenhuis, Doetinchem
  - Leiden University Medical Center, Leiden
  - Erasmus MC, Rotterdam

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kok S, Schoonhoven L, Vernooij LM, Reitsma JB, Verstraten C, Metzelthin SF, Bleijenberg N, de Man-van Ginkel JM. The effectiveness of Function Focused Care among patients acutely admitted to hospital: A stepped wedge cluster trial. Int J Nurs Stud. 2024 Dec;160:104893. doi: 10.1016/j.ijnurstu.2024.104893. Epub 2024 Sep 4. PMID 39321557
- [Background] Kok S, de Man-van Ginkel JM, Verstraten C, Resnick B, Metzelthin SF, Bleijenberg N, Schoonhoven L. Function focused care in hospital: A mixed-method feasibility study. Int J Nurs Stud Adv. 2021 Sep 29;3:100045. doi: 10.1016/j.ijnsa.2021.100045. eCollection 2021 Nov. PMID 38746732